CLINICAL TRIAL: NCT07024004
Title: Effects of Active Exergames Program on Muscle Strength, Lower Limb Muscle Mass and Physical Fitness in Older Adults at Risk of Falls
Brief Title: Active Exergames Program in Older Adults at Risk of Falls
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Catolica Silva Henriquez (Other)
Collaborators: Agencia Nacional de Investigacion y Desarrollo, ANID (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANID-NAM N°NAM24I0019
Record Dates: First submitted 2025-04-05; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Risk of Falls
Keywords: Exergames; Virtual Reality Exercise; Older Adults; Fall Prevention

STUDY DESIGN:
Intervention Model Description: Parallel Assignment:
  This study uses a parallel assignment model, where participants are randomly assigned to one of two groups:
  Group 1 receives a combined intervention of exergame-based exercise and conventional physical therapy.
  Group 2 receives conventional physical therapy alone.
  The interventions are conducted simultaneously over a 12-week period, 2 sessions per week of one hour each, and comparisons are made between and within groups to evaluate outcomes such as lower limb strength, muscle quality, and physical function.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exergame-Based Exercise + Conventional Physical Therapy group (Experimental): Participants in this group will receive a combined intervention that includes multicomponent physical exercise and training using exergames (specifically Ring Fit Adventure on the Nintendo Switch). The sessions target strength, balance, and aerobic capacity and will be delivered twice a week for 12 weeks in senior care centers.
  Interventions: Behavioral: Exergame-Based Exercise + Conventional Physical Therapy
- Conventional Physical Therapy Group (Active Comparator): Participants in this group will receive a standard multicomponent physical exercise program including aerobic, strength, balance, and flexibility exercises, delivered twice a week for 12 weeks in senior care centers. No exergames or virtual reality components will be included in this intervention.
  Interventions: Behavioral: Conventional Physical Therapy

INTERVENTIONS:
Behavioral: Exergame-Based Exercise + Conventional Physical Therapy — Participants in this group will engage in a combined intervention consisting of:
  Multicomponent physical exercise (aerobic, strength, balance, and flexibility), delivered twice per week for 12 weeks.
  Exergames training using the Nintendo Switch console and Ring Fit Adventure game. Sessions include warm-up, gameplay involving full-body movements (e.g., squats, running, balance tasks), and cooldown.
  Sessions are adapted to individual physical capacities and supervised by a trained kinesiologist.
  The intensity is monitored using the Borg Scale, following ACSM guidelines.
  Arms: Exergame-Based Exercise + Conventional Physical Therapy group
Behavioral: Conventional Physical Therapy — Participants in this group will receive a standard multicomponent physical exercise program consisting of:
  Exercises for aerobic capacity, strength, balance, and flexibility.
  Delivered in-person twice per week for 12 weeks at senior care centers.
  Sessions include warm-up (5-10 min), main activity (30-40 min), and cooldown (5-10 min).
  Intensity is controlled using the Borg Scale and monitored by a supervising kinesiologist.
  Arms: Conventional Physical Therapy Group

SUMMARY:
The goal of this randomized clinical trial is to analyze the effectiveness of a physical exercise program based on exergames combined with conventional physical therapy, compared to a conventional physical exercise program alone, in improving lower limb strength, muscle quality, and physical capacity in older adults at risk of falling. The main questions it aims to answer are:

Does a combined exergame and conventional exercise program improve functional capacity in older adults at risk of falling more than traditional exercise alone? Does the intervention improve lower limb strength and muscle quality more effectively than conventional exercise alone?

Researchers will compare a group receiving exergame-based exercise combined with conventional therapy to a group receiving conventional physical exercise only to see if the addition of exergames enhances functional outcomes and muscle performance.

Participants will:

* Undergo baseline and post-intervention assessments of lower limb strength, muscle quality, and physical capacity.
* Participate in a structured physical exercise program.
* In the intervention group, perform exergame-based exercises using virtual reality gaming systems such as Nintendo Switch (Ring Fit Adventure).
* Engage in sessions for several weeks, with consistent frequency and intensity depending on the group allocation.

DETAILED DESCRIPTION:
Falls in older adults have been associated with a decrease in physical activity, the level of functionality and an increase in dependency. Furthermore, falls and their consequences are one of the main causes of mortality among older people. Falls are more frequent in women, in people over 75 years of age and with sensory deficits.

Currently, there are promising and novel solutions to prevent and/or avoid the repetition of falls; Among them, the use of active exergames stands out. Active exergames can be developed in health, community, sports centers or in a homeroom individually or in groups using a screen through video games that involve the movement of the whole body, like the real world with or without the use of a controller that allows you to execute movements in a small space and interact with the game scenario. They have been shown to be useful for improving balance and physical condition in people of different ages and health conditions, but there is little evidence of studies that analyze the effects of this therapeutic strategy in older adults at risk of falling.

Active exergames are a novel, simple, motivating, and easy-to-implement treatment option to promote healthy aging and prevent the risk of falls in older people. Therefore, it has the potential to become, in the short term, a therapeutic strategy for mass use, with high adherence and low cost in health centers.

Exergames have an affordable cost, with a wide variety of games and are easy to use, therefore it is increasingly accepted by different types of patients as a therapeutic strategy.

The evidence indicates that, both programs are expected to improve the primary and secondary outcomes proposed in this project. Additionally, older adults who execute an active exergame program are expected to have better performance compared to a conventional physiotherapy program in the main outcome and the secondary outcomes analyzed. It is expected to promote the use of active exergames by rehabilitation professionals in primary health care centers to prevent falls in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or older
* Both sexes eligible
* Attendees of SENAMA day centers (senior care centers) in the Metropolitan Region of Santiago, Chile.
* Mini-Mental State Examination (MMSE) score > 14
* Barthel Index score > 60 (indicating moderate to good functional independence)
* No self-reported medical contraindications for physical exercise
* Ability to walk independently (with or without assistive devices)
* Provided written informed consent

Exclusion Criteria:

* Recent bone fractures or acute myocardial infarction
* Severe cardiovascular or respiratory conditions
* Uncontrolled hypertension or diabetes mellitus
* Cognitive or sensory impairments that limit instruction comprehension
* Participation in other exercise programs during the study period
* Inability to attend at least 80% of the intervention sessions

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Risk of fall | Baseline and 12 weeks post-intervention
  Fall risk will be evaluated using the Downton Fall Risk Index (DFRI), a 5-item composite score based on prior falls, medication, sensory deficits, mental state, and mobility. A total score >3 indicates high fall risk.
Functional Independence | Baseline and 12 weeks post-intervention
  Functional independence will be measured with FIM scale, it consists of 18 items that assess both motor and cognitive skills, and is scored on a 7-level scale, where 1 indicates total dependence and 7 complete independence.
Center of Pressure (COP) | Baseline and 12 weeks post-intervention
  Posturography, which records center of pressure displacement while standing on a stable platform.
Dynamic balance | Baseline and 12 weeks post-intervention
  Dynamic balance is measured with the Timed Up and Go (TUG) test, which evaluates the time in seconds that a participant takes to rise from a chair, walk 3 meters, turn, return, and sit down again.
Static balance | Baseline and 12 weeks post-intervention
  Single-Leg Stance Test (Unipedal Stance Test), where participants must maintain balance on one leg for at least 5 seconds.
Aerobic capacity | Baseline and 12 weeks post-intervention
  Aerobic capacity is assessed by the 2-Minute Walk Test, which measures the total distance (in meters) covered at a self-selected walking pace within 2 minutes on a flat surface.

SECONDARY OUTCOMES:
body composition | Baseline and 12 weeks post-intervention
  Segmental muscle mass of the lower limbs will be assessed using a bioelectrical impedance analyzer (InBody 270). The participant stands barefoot and holds electrodes as the device estimates muscle mass.
Handgrip strength | Baseline and 12 weeks post-intervention
  handgrip strength will be assessed bilaterally in a seated position using a handheld dynamometer with the elbow at 90° flexion. The highest value from three attempts will be recorded (in kilograms).
Lower Limb Muscle Strength | Baseline and 12 weeks post-intervention
  Strength of the lower limbs will be evaluated using the Five Times Sit-to-Stand Test (FTSST). Participants are asked to sit and stand from a chair five times as quickly as possible, with arms crossed over the chest. The time taken (in seconds) will be recorded.
Intramuscular Fat Infiltration | Baseline and 12 weeks post-intervention
  Muscle echogenicity will be measured via ultrasound (transversal view of the quadriceps). Images will be analyzed using ImageJ software to calculate grayscale intensity (0-255 arbitrary units), which reflects intramuscular fat content.
Muscle Architecture | Baseline and 12 weeks post-intervention
  Muscle architecture (muscle thickness, pennation angle, fascicle length) of the quadriceps will be evaluated through ultrasound imaging. These anatomical variables will be analyzed using ImageJ software.

CONTACTS AND LOCATIONS:
Overall Officials: Paloma Lillo Urzúa, MSc, Principal Investigator — Universidad Católica Silva Henríquez
Locations (1):
- Universidad Católica Silva Henríquez, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No
The informed consent signed by participants does not include authorization to share individual data publicly or with third parties.

REFERENCES:
- [Background] Deng N, Soh KG, Abdullah BB, Tan H, Huang D. Active video games for improving health-related physical fitness in older adults: a systematic review and meta-analysis. Front Public Health. 2024 Apr 17;12:1345244. doi: 10.3389/fpubh.2024.1345244. eCollection 2024. PMID 38694976
- [Background] Hernandez-Martinez J, Ramos-Espinoza F, Munoz-Vasquez C, Guzman-Munoz E, Herrera-Valenzuela T, Branco BHM, Castillo-Cerda M, Valdes-Badilla P. Effects of active exergames on physical performance in older people: an overview of systematic reviews and meta-analysis. Front Public Health. 2024 Apr 9;12:1250299. doi: 10.3389/fpubh.2024.1250299. eCollection 2024. PMID 38655514
- [Background] Taylor LM, Kerse N, Frakking T, Maddison R. Active Video Games for Improving Physical Performance Measures in Older People: A Meta-analysis. J Geriatr Phys Ther. 2018 Apr/Jun;41(2):108-123. doi: 10.1519/JPT.0000000000000078. PMID 26974212
- [Background] Suleiman-Martos N, Garcia-Lara R, Albendin-Garcia L, Romero-Bejar JL, Canadas-De La Fuente GA, Monsalve-Reyes C, Gomez-Urquiza JL. Effects of active video games on physical function in independent community-dwelling older adults: A systematic review and meta-analysis. J Adv Nurs. 2022 May;78(5):1228-1244. doi: 10.1111/jan.15138. Epub 2021 Dec 21. PMID 34935178
- [Derived] Lillo-Urzua P, Ugarte-Llanten J, Carreno-Zilmann G, Vidal-Seguel N, Guede-Rojas F, Cuenca-Garcia M, Cigarroa I. E-ACTIVE AGING study protocol: Evaluating an exergame-based and multicomponent exercise program for community-dwelling older adults at risk of falling. Front Physiol. 2025 Dec 3;16:1691454. doi: 10.3389/fphys.2025.1691454. eCollection 2025. PMID 41415308